CLINICAL TRIAL: NCT01152749
Title: Bioequivalence Between an Oral Nicotine Replacement Product and Nicorette® Gum. A Study in Healthy Smokers.
Brief Title: Bioequivalence Between an Oral Nicotine Replacement Product and Nicorette® Gum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICTDP1075; 2009-010633-44 (EudraCT Number)
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Tobacco Dependence
Keywords: Smoking Cessation; Nicotine pharmacokinetics
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Nicotine; Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- UNG-GC-2 (Experimental): 2 mg experimental NRT product
  Interventions: Drug: Nicotine
- UNG-GC-4 (Experimental): 4 mg experimental NRT product
  Interventions: Drug: Nicotine
- Nicorette® Gum-2 (Active Comparator): 2 mg Nicorette® Gum
  Interventions: Drug: Nicotine Gum
- Nicorette® Gum-4 (Active Comparator): 4 mg Nicorette® Gum
  Interventions: Drug: Nicotine Gum

INTERVENTIONS:
Drug: Nicotine — Single-dose of new NRT product
  Other Names: Nicotine NRT / not yet marketed
  Arms: UNG-GC-2; UNG-GC-4
Drug: Nicotine Gum — Single-dose of marketed nicotine gum
  Other Names: Nicorette® Gum
  Arms: Nicorette® Gum-2; Nicorette® Gum-4

SUMMARY:
This study examines the bioequivalence between an oral nicotine replacement product and Nicorette® gum.

DETAILED DESCRIPTION:
The study is a single-dose, randomized, crossover study with 76 subjects (all subjects will receive all treatments). The investigational products will be given as single doses at separate treatment visits. Periods without Nicotine Replacement Therapy (NRT), lasting for at least 36 hours, will separate treatment visits. Blood for pharmacokinetic analyses will be drawn before and at 5, 10, 15, 20, 30, 45, and 60 minutes, as well as at 1.5, 2, 4, 6, 8, and 10 hours after start of product administration. Used gums will be collected and analyzed to determine the amount of remaining nicotine. Subjects will also be monitored to capture any adverse events that may occur.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, smoking at least 10 cigarettes daily during at least one year preceding inclusion and body mass index (BMI) between 17.5 and 30.0 kg/m2.
* Female participants of child-bearing potential are required to use a medically acceptable means of birth control.
* A personally signed and dated informed consent document, indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Pregnancy, lactation or intended pregnancy.
* Treatment with an investigational product or donation or loss of blood within 3 month preceding the first dose of study medication.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2009-12; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic measurements | Baseline and during 10 hours after product administration
  Pharmacokinetic measurements including:
  * the maximum observed nicotine concentration in plasma (Cmax)
  * the area under the plasma concentration-vs.-time curve until the last measurable concentration (AUCt)
  * the area under the plasma concentration-vs.-time curve until infinity (AUC∞)

SECONDARY OUTCOMES:
tmax | Baseline and during 10 hours after product administration
  The time of occurrence of Cmax following product administration
Lamda z | Baseline and during 10 hours after product administration
  The terminal nicotine elimination rate constant (λz)
Released amount of nicotine | After 30 minutes of chewing
  The amount of nicotine released from gums during 30 minutes' chewing.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- McNeil AB Clinical Pharmacology R&D, Lund, Sweden